CLINICAL TRIAL: NCT05845060
Title: Reliabılıty,Validity Of The Turkish Version Of The Lumbar Spine Surgery Exceptations
Brief Title: Lumbar Spine Surgery Exceptations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Aydın Sinan Apaydin, Director, Karabuk University
Other Study IDs: KarabukUniversity
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Low back pain is one of the most common reasons for applying to health institutions. Low back pain seriously affects the lives of patients and causes great financial losses. Surgical treatments have an important place in the treatment of pain due to lumbar spine pathologies. Although success in lumbar spine surgery depends on many factors, it has been reported that one of the most important of these factors is patient expectations. In order for patients and doctors to have the same priorities and meet the same realistic goals, it is necessary to understand what patients expect. Many studies have attempted to measure patients' expectations for lumbar spine treatment; however, most of them are unapproved, valid and unreliable scales. Lumbar spine surgery expectations scale was created by Mancuso et al. in 2013 to learn the expectations of patients in lumbar spine surgery. It has been found that the scale has high validity and reliability values and it has been observed that it is frequently used in clinics and researches. In our country, there is no valid and reliable scale that questions the expectations of patients from lumbar surgery. As a result of this study, it is planned to introduce a valid and reliable scale adapted into Turkish, which can question the expectations of patients from a lumbar surgery.

DETAILED DESCRIPTION:
Low back pain is one of the most common reasons for applying to health institutions. Low back pain seriously affects the lives of patients and causes great financial losses. Surgical treatments have an important place in the treatment of pain due to lumbar spine pathologies. Although success in lumbar spine surgery depends on many factors, it has been reported that one of the most important of these factors is patient expectations. In order for patients and doctors to have the same priorities and meet the same realistic goals, it is necessary to understand what patients expect. Many studies have attempted to measure patients' expectations for lumbar spine treatment; however, most of them are unapproved, valid and unreliable scales. Lumbar spine surgery expectations scale was created by Mancuso et al. in 2013 to learn the expectations of patients in lumbar spine surgery. It has been found that the scale has high validity and reliability values and it has been observed that it is frequently used in clinics and researches. In our country, there is no valid and reliable scale that questions the expectations of patients from lumbar surgery. As a result of this study, it is planned to introduce a valid and reliable scale adapted into Turkish, which can question the expectations of patients from a lumbar surgery.

Developing the scale in order to carry out the Turkish validity and reliability study of the Lumbar Spine Surgery Expectations scale and to confirm that the Turkish validity and reliability of the questionnaire was not done by another researcher, Prof. Dr. Mancuso Carol was contacted via e-mail and necessary permissions were obtained from him. The scale will be translated into Turkish by the study team after the approval of the ethical committee that there is no ethical objection to the conduct of the study. For this purpose, three researchers whose mother tongue is Turkish and fluent in English will separately translate the scale into Turkish, and then the final version of the scale will be obtained by three researchers. Physicians and physiotherapists working at KBU Training and Research Hospital will be asked to read the final version of the scale and evaluate the items in a way that is easy to understand and difficult to understand. Items that are stated to be difficult to understand will be reviewed. The scale items, whose intelligibility has been determined, will be translated into English by a translator whose native language is English and who is fluent in Turkish. The developer of the scale questionnaire translated into English, Prof. Dr. Mancuso will be sent to Carol and asked to evaluate whether there is consistency in meaning between the original scale and the translated scale. If the items are consistent, the Turkish version of the scale will be determined and it will be applied to patients who are planned for lumbar spine surgery. Together with the developed scale and Quebeck Waist Disability Scale, it will be applied to the patients by face-to-face method. In this way, the consistency of the developed scale with similar questionnaires that were previously reported to be valid will be examined. In order to determine the reliability of the scale, it will be applied again to the participants who agreed to fill in the questionnaire again one week later. The consistency of the scale will be determined by the data of the participants with the first and second scale scores.

ELIGIBILITY:
Inclusion Criteria:

1. 18 -65 years old
2. To be able to read and write Turkish
3. To have lumbar spine surgery planned by neurosurgery or orthopedist

Exclusion Criteria:

1. Being scheduled for revision surgery
2. Having a cognitive deficit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample of this study will consist of volunteer patients who applied to the Neurosurgery outpatient clinic of Karabuk University Training and Research Hospital and who were at the surgical level due to chronic low back pain.
Sampling Method: Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Lombar Spine Surgery Expectitaions | 10 minutes
  Lumbar spine surgery expectations scale was created by Mancuso et al. in 2013 to learn the expectations of patients in lumbar spine surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Gunes, MSC, Principal Investigator — Karabük University; Metehan Yana, Phd, Principal Investigator — Karabük University; Ismail Saracoglu, Phd, Principal Investigator — Kutahya Health Science University; Cihan Caner Aksoy, Phd, Principal Investigator — Kutahya Health Science University
Locations (1):
- Karabuk University, Karabük, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Mancuso, C. A., Cammisa, F. P., Sama, A. A., Hughes, A. P., Ghomrawi, H. M., & Girardi, F. P. (2013). Development and testing of an expectations survey for patients undergoing lumbar spine surgery. JBJS, 95(19), 1793-1800. 2. Aoude, A., Litowski, M., Aldebeyan, S., Fisher, C., Hall, H., Manson, N., ... & Paquet, J. (2020). A Comparison of Patient and Surgeon Expectations of Spine Surgical Outcomes. Global Spine Journal, 2192568220907603. 3. Nepomuceno, E., Silveira, R. C. D. C. P., Dessotte, C. A. M., Furuya, R. K., Arantes, E. D. C., Cunha, D. C. P. T. D., & Dantas, R. A. S. (2016). Instruments used in the assessment of expectation toward a spine surgery: an integrative review. Revista da Escola de Enfermagem da USP, 50(4), 658-666.